CLINICAL TRIAL: NCT04969094
Title: Reducing Fall Risk With the Use of Neuromuscular Electrical Stimulation to Maximize the Hip Abductor Muscles in Older Veterans
Brief Title: Reducing Fall Risk With NMES
Acronym: NMES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E3484-R; RX003484 (Other Grant/Funding Number: Veteran Affairs Rehabilitation R&D Service)
Record Dates: First submitted 2021-07-07; First posted 2021-07-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Falls
Keywords: Fall

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES + MMBI (Experimental): Neuromuscular electrical stimulation applied to hip abductors along with participation in a multi-modality balance intervention
  Interventions: Other: Neuromuscular electrical stimulation (NMES); Other: Multi-Modality Balance Intervention (MMBI)
- MMBI (Active Comparator): Participation in a multi-modality balance intervention
  Interventions: Other: Multi-Modality Balance Intervention (MMBI)

INTERVENTIONS:
Other: Neuromuscular electrical stimulation (NMES) — Participants will receive NMES to the hip abductors while performing strength training 3 times per week for 3-months
  Arms: NMES + MMBI
Other: Multi-Modality Balance Intervention (MMBI) — Participants will attend a group balance class that focuses on movement and obstacle negotiation 3 times per week for 3-months

SUMMARY:
Falls are dangerous leading to injuries, hospital admissions and even death. Fall prevention is a priority but effective programs only reduce falls by 30%. Weak hip muscles may be one reasons individuals experience a loss of balance. However individuals who have weak hip muscles may be unable to exercise at sufficient intensities to improve their hip muscle strength. The purpose of this study is to utilize a common physical therapy method, neuromuscular electrical stimulation (NMES), on the hip muscles to improve hip muscle strength and improve balance. The new program focuses on using NMES during a resistance training program along with exercise to improve standing balance, walking and stepping over objects. This study will test the additive effect of NMES applied to the hip muscles during a balance and strengthening program to improve balance and mobility, and ultimately reduce the risk of falls in older Veterans at high risk for falls.

DETAILED DESCRIPTION:
Falls are a leading cause of disability in older adults. Decreased lower extremity muscle mass and strength contribute to balance and mobility limitations. More recent work also suggests that in addition to the traditional targets of muscle mass of the thigh and leg muscles, dysfunction of the hip abductors may contribute to balance and mobility limitations resulting in increased fall risk. Older adults with impaired hip abductor muscles demonstrate increased amounts of intramuscular fat (IMAT) in and around the muscles, decreased hip abductor strength, lower balance scores, increased gait variability (a predictor of future falls), and poor stepping mechanics when recovering from a balance perturbation. Increased IMAT and muscle dysfunction of the hip abductors may contribute to poor hip abductor muscle recruitment and make changing these muscle during a traditional intervention difficult. Neuromuscular electrical stimulation (NMES) is one method to improve muscle mass, strength and quality in older adults, but has not traditionally been used on the hip abductors. The investigator's central hypothesis is that the addition of NMES applied to the primary hip abductors during a multimodality balance intervention (MMBI) will result in greater reduction in fall risk and larger improvements in muscle and mobility function than MMBI alone. The investigators will test this hypothesis with the following specific aims:

Aim 1: To determine the 3-month effects of a multimodality balance intervention with and without NMES on fall risk.

Aim 2: To examine the 3-month effects of a multimodality balance intervention with and without NMES on functional outcomes including muscle function and composition.

Aim 3: To evaluate the retention of balance, muscle changes and reduced falls after a multimodality balance intervention with and without NMES

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* At risk for falls

Exclusion Criteria:

* Poorly controlled hypertension
* Home oxygen use
* Contraindications to resistance exercise
* Contraindications for NMES use
* Dementia
* Other medical condition precluding patient participation in this study as per medical judgment of study team

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Balance | 3-months
  The four-square step test will be used as a measure of balance. The change in the amount of time it takes to complete the four-square step test comparing pre and post-intervention.
Isometric Hip Abductor Strength | 3-months
  A measure of the maximal isometric muscle strength produced in hip abductor muscles will be assessed with a biodex device. Pre-test levels will be compared to post-intervention levels.

SECONDARY OUTCOMES:
Mobility | 3-months
  The modified physical performance test is a mobility measure that utilizes 9 tasks scored 0-4 (total possible score 36) to determine functional status. Pre-test scores will be compared to post intervention test scores.
Muscle composition | 3-months
  A measure of the amount of muscle and fat in the muscle using a CT scan of the hips. Pre-test levels will be compared to post intervention levels
Balance | 12-months after Exercise completion
  The change in the amount of time it takes to complete the four-square step test comparing post-intervention to 12-months after the cessation of exercise.
Isometric Hip Abductor Strength | 12-months after Exercise completion
  A measure of the maximal isometric muscle strength produced in hip abductor muscles will be assessed with a biodex device.. Post-intervention levels will be compared to 12 months after the cessation of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Odessa R. Addison, PhD DPT, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedman B, Beamer BA, Beans J, Gray V, Alon G, Ryan A, Katzel LI, Sorkin JD, Addison O. Neuromuscular Electrical Stimulation to Maximize Hip Abductor Strength and Reduce Fall Risk in Older Veterans: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 May 1;14:e68082. doi: 10.2196/68082. PMID 40312027